CLINICAL TRIAL: NCT03042416
Title: 18F-DOPA PET Imaging: an Evaluation of Biodistribution and Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00055342
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Congenital Hyperinsulinism; Neuroblastoma; Neuroendocrine Tumors; Parkinson Disease; Brain Glioma
Keywords: 18F-DOPA PET/CT
MeSH Terms: conditions — Congenital Hyperinsulinism; Neuroblastoma; Neuroendocrine Tumors; Parkinson Disease | interventions — fluorodopa F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-DOPA scan (Experimental): 18F-DOPA (4 MBq/kg, minimum 110 MBq, maximum 600 MBq) intravenous. Single-dose 20-80 minutes prior to PET/CT scan of brain or whole body (depending on specific imaging protocol for patient).
  Interventions: Drug: 18F-DOPA

INTERVENTIONS:
Drug: 18F-DOPA — 18F-DOPA intravenous injection single dose

SUMMARY:
Single centre prospective cohort phase III study of 18F-DOPA PET/CT imaging in specific patient populations:

1. Pediatric patients with congenital hyperinsulinism
2. Pediatric patients with neuroblastoma
3. Pediatric or Adult patients with suspected extra-pancreatic neuroendocrine tumor
4. Adult patients with a clinical suspicion of Parkinson's disease
5. Pediatric or Adult patients with primary brain tumors

This study will evaluate the biodistribution and safety of 18F-DOPA produced at the Edmonton PET Centre.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pediatric patients (less than 17 years old) with congenital hyperinsulinism
* 2. Pediatric patients (less than 17 years old) with neuroblastoma
* 3. Pediatric patients (less than 17 years old) or Adult patients (17 or older) with known or clinically suspected neuroendocrine tumor outside of the pancreas
* 4. Adult patients (17 or older) with a clinical suspicion of Parkinson's disease.
* 5. Pediatric (less than 17 years old) or Adult patients (17 or older) with primary brain tumors

Exclusion Criteria:

* Unable to obtain consent
* Weight > 250 kg (weight limitation of PET/CT scanner)
* Adult patients unable to lie flat for 20-30 minutes to complete the PET/CT scan
* Young pediatric patients (less than 10 years old) who are unable to lie flat for 20-30 minutes and for whom clinical sedation is contraindicated (as determined by a pediatric anaesthesiologist)
* Pregnancy
* Lack of intravenous access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Immediate safety evaluation | Within 1 hour of injection
  Clinical screen for adverse reactions to 18F-DOPA injection

SECONDARY OUTCOMES:
Delayed safety evaluation | 10-14 days after injection
  A telephone survey to evaluate for delayed adverse reactions to 18F-DOPA injection
Delayed safety evaluation - referring physician | 6 months after injection
  Questionnaire for referring physician to screen for adverse reactions to 18F-DOPA injection
Biodistribution: scan interpreter will evaluate the distribution of tracer and comment if expected | Within 3 days after injection
  Scan interpreter will evaluate the distribution of tracer and comment if expected
Perceived clinical benefit | 6 months after injection
  Questionnaire for referring physician to assess perceived clinical benefit of scan

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan T Abele, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No